CLINICAL TRIAL: NCT06337201
Title: A Digital Life Story to Support Person-centred Care for Older Adults With Dementia: Healthcare Professionals' Perspectives
Brief Title: A Digital Life Story to Support Person-centred Care for Older Adults With Dementia Perspectives
Status: Recruiting | Type: Observational
Sponsor: Blekinge Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: BTH-6.1.1-0138-2023
Record Dates: First submitted 2024-01-29; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Cognitive Impairment; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare professionals working in daycare center and residential care.
  Interventions: Device: Test of the application Min Memoria

INTERVENTIONS:
Device: Test of the application Min Memoria — Focus group interviews will be conducted to reach healthcare professionals' experiences using a written life story in daily care. Then, the information from the written life story will be transferred to the application, and the healthcare professionals will test a digital life story (the application) in daily care instead. Observation studies will be conducted to observe the use of the digital life story. What can be seen in the communication and the interaction, and in what situations is the digital life story used?

SUMMARY:
Person-centred care can be supported when healthcare professionals access and actively use the information recorded in a life story. Active use of the life story can create security for a person with dementia and their carers. The written life story describes the person and their life experiences, which can define the person's identity. National guidelines for care and nursing in dementia and Blekinge's regional guidelines emphasise the importance of care and nursing for people with dementia, which should be given with a person-centred approach, where the life story becomes a tool for healthcare professionals. Research shows that a life story can be designed in several ways. For example, in book form, as a brochure, collage, memory box or electronically. The life story is also intended as a tool for healthcare professionals to create security and facilitate communication with the individual. As more and more older adults are using computers and tablets as assistive devices, and it is also becoming more common for healthcare professionals to use, for example, tablets as assistive devices in nursing care, the life story could be shared in digital form as an application and become a living document.

Overall aim: To test an application for the life story with the intention of supporting person-centred care for older adults with dementia and to test whether the application can replace the written completion document. Study I: Exploring the research area of the life story in digital form. Study II: Focus group interviews with healthcare professionals. Study III: Test the application, Min Memoria. Study IV: Observations on the use of the application.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals using a life story in daily care.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals working in daycare center and residential care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Healthcare professionals' experiences using a written life story in the daily care of older adults with dementia | From October 2023 - August 2024
  Focus group interviews
Data on the use of a digital life story tool. | September 2024 - August 2025
  Explore the usability, accessibility and positive and negative effects on daily care. Data will be collected through a survey with healthcare professionals (participants).
Observation when using a digital life story | September 2025 - December 2026
  Data will be collected through non-participant observations. Observing communication and interactions between the healthcare professionals and the older adults when using the digital tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Blekinge Institute of Technology, Karlskrona, Blekinge County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The data supporting this study's findings will be available on request from the corresponding author (Helén Dellkvist). The data are not publicly available due to privacy or ethical restrictions.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: From when each sub-study is publiced and onwards.